| Official Title Randomized, placebo-controlled, phase II trial e ustekinumab for prevention of graft vs. host | |
|---|---|
| | disease after allogeneic hematopoietic cell transplantation |
| NCT Number | NCT04572815 |
| <b>Document Type</b> | Informed Consent Form |
| <b>Document Date</b> | 5/3/2023 |

# Fred Hutchinson Cancer Center Moffitt Cancer Center

# Consent to take part in a research study:

# Randomized, placebo-controlled, phase II trial examining ustekinumab for prevention of graft vs. host disease after allogeneic hematopoietic cell transplantation

Principal Investigator: Stephanie Lee, MD, MPH. University of Washington; Fred

Hutchinson Cancer Center. 206-667-5160

# Emergency number (24 hours): (206) 598-8902

Ask to page the Long-Term Follow-Up Attending

# Important things to know about this study.

You are invited to participate in a research study. The purpose of this research is determine whether adding ustekinumab (Stelara<sup>TM</sup>) to the existing medication regimen of tacrolimus and methotrexate will help reduce the risk of developing graft-vs-host disease (GVHD) better than tacrolimus and methotrexate alone. GVHD is a complication of an allogeneic transplant, a transplant using blood cells that come from someone other than yourself (a donor).

People who agree to join the study will be asked to attend 26 visits over about two years. Most of the study visits occur in the first 4 months. The study involves frequent physical exams, blood draws, questionnaires, and other assessments.

We do not know if ustekinumab would help prevent GVHD, and it could even make your condition/disease worse. Ustekinumab could cause side effects such as headaches, dizziness, and redness at the study drug injection site, as described below in this form.

You do not have to join this study. You can choose to receive standard methods to prevent GVHD instead of participating in this study. We will give you details about the purposes, procedures, risks and possible benefits related to this study. We will explain other choices that you have. We will also give you any other information that you need in order to make an informed decision about joining this study.

Following is a more complete description of this study. Please read this description carefully. You can ask any questions you want to help you decide whether to join the study. If you join this study, we will give you a signed copy of this form to keep for future reference.

# We invite you to join this research study.

We invite you to join this research study because you are a candidate for allogeneic transplant, and therefore you will be at risk for the complication of transplant called graft vs. host disease (GVHD). Up to 116 people at 4 transplant centers will join this study.

Research is not the same as treatment or medical care. The purpose of a research study is to answer scientific questions.

You do not have to be in the study. You are free to say "yes" or "no", or to drop out after joining. If you say "no," you would have no penalty or loss of benefits. Whatever you decide, your regular medical care would not change.

# Why are we doing this study?

We are doing this study to determine whether adding ustekinumab to the existing medication regimen of tacrolimus and methotrexate will reduce the risk of developing GVHD after transplant. GVHD is a disease caused by an immune reaction of donor cells against patient tissues. Many organs of the body (skin, eyes, mouth, hair, liver, gastrointestinal tract, lungs and joints) may be damaged by this disease. If GVHD becomes severe, it can be disabling or can lead to death. Some of the patients who survive may be severely disabled from progressive hardening of the skin, tightening (contractures) of the joints, drying of the eyes and weight loss. Medication must be given for prevention of GVHD.

Tacrolimus and methotrexate are two standard medications used to prevent GVHD or reduce the severity of GVHD after allogeneic hematopoietic stem cell transplant. This study will compare the standard medications (tacrolimus and methotrexate) to tacrolimus, methotrexate, and ustekinumab.

Ustekinumab is FDA-approved for the treatment of psoriasis and Crohn's disease. Psoriasis is a common skin condition that causes skin redness and irritation. Ustekinumab is not FDA-approved for the prevention of GVHD. However, ustekinumab has been studied in several human conditions (such as multiple sclerosis, inflammatory bowel disease, and others) that have similarity to GVHD. Specifically, ustekinumab targets signals that drive unwanted immune responses that underlie the problem of GVHD. Therefore, there is reason to suspect that it could be helpful in preventing GVHD. Ustekinumab, an investigational treatment for GVHD, has been previously given as GVHD prevention in a prior clinical trial of 30 patients total. This current larger study will more completely test whether this is helpful in preventing GVHD.

There are 2 groups of participants in this study. We will give different treatments to different groups and compare the results. This is how we hope to find out if ustekinumab helps to prevent GVHD.

Group 1: Tacrolimus and methotrexate plus ustekinumab

• Group 2: Tacrolimus and methotrexate plus placebo

All patients in this study will receive tacrolimus and methotrexate. If you join this study, you would also receive ustekinumab or a placebo. A placebo does not have the active ingredients in ustekinumab. A computer program will be used to decide which treatment you receive. If you join this study, you would not be allowed to choose the treatment. You would have a 1-in-2 chance of receiving ustekinumab. Neither you nor your doctor will know to which group you have been assigned.

# What research tests, procedures, and treatments are done in this study?

Before starting the study drug, you would need to complete a screening visit. If you complete the screening visit and enroll in the study, you will have study visits in the hospital, office, or clinic at least once a week for the first 100 days post-transplant. After Day +100, you will return for follow-up visits at 4, 6, 9, 12, 18, and 24 months. A full schedule of study visits is on page 5 of this consent form.

If you decide to join this study, we will do these tests and procedures:

- Questionnaires We would ask you to fill out five questionnaires—one before your transplant, one about 100 days after your transplant, and three more in the follow-up period (6 months, 1 year, and 2 years post-transplant). Each questionnaire includes questions about your GVHD symptoms, physical and mental health, and your quality of life. Some of the questions may be sensitive. Questions that make you feel uncomfortable would not have to be answered.
- Clinical Assessment You will have a physical exam at most study visits, and we will pay special attention to any signs or symptoms of GVHD that you may be having. A member of the study team will fill out a form about your GVHD. We will collect your vital signs, height, and weight. You will be watched very closely by your doctor for infections, recurrence of your disease and for any side effects.
- Study Drug (ustekinumab or placebo) The study drug will be given by vein or as a shot under your skin. The first dose will be given in your vein up to three days before you start transplant conditioning therapy. Additional doses will be given as a shot about every 8 weeks after transplant (Day +50, Day +100, Day +160). You will receive 4 doses of the study drug. The placebo will be given as a sterile saline (identical volume to that of ustekinumab) with no active medicine.
- Tacrolimus Tacrolimus will be started before your transplant. It may be administered orally or as an intravenous (IV) infusion. If you receive it intravenously, we will change the administration of tacrolimus to a pill form as soon as possible after transplant. The dose of tacrolimus will be adjusted depending on side effects and the level of tacrolimus in your blood. In some cases, we may hold the dose of tacrolimus. It is planned that tacrolimus will

be given for about 180 days after transplant, although it often continues beyond this time, particularly if GVHD occurs. To measure the level of tacrolimus in your blood, we will draw blood from the catheter (tube) or port in your chest, or from your arm. This will be done once a week, and possibly more often. The amount of blood needed is less than one teaspoon.

- Methotrexate Methotrexate will be given as an IV infusion on days 1, 3, 6 and 11 after transplant. Depending on side effects and your clinical condition, the dose of methotrexate might be reduced or not given. After you are given methotrexate, we may check the level of this medication in your blood. Again, this blood will be drawn from your catheter, port, or vein. The amount of blood needed is less than one teaspoon.
- Clinical labs We will do blood tests to check for GVHD and overall health. Most of the time, these labs will be done as part of your normal medical care.
- Research blood samples By taking part in this study, you would also have additional research blood samples obtained that are not part of standard of care. With these blood samples, we will determine how the study therapy influences certain cells and other signals within your immune system. We will collect 18 mL (about 1 1/2 tablespoons) four times for research. We will collect 60 mL (about 4 tablespoons) seven times for research.
- Research bone marrow samples If a bone marrow procedure is performed for clinical samples, you may be asked to give an extra 1-2 teaspoons (5-10ml) of liquid bone marrow sample. Withdrawal of the extra marrow may cause 5-10 seconds of additional temporary discomfort. We will make every effort to collect the sample using the same point of entrance for the needle. Very rarely would we need to reposition the needle to collect the research sample.
- **Pregnancy test** If you are a woman of childbearing potential, we will do a blood test to check for pregnancy before you begin taking the study drug.

# Study visits

# **Schedule of Study Visits and Procedures**

# **Study Procedures**

| | , | Study 1 1000du103 | | | | | |
|---|---|---|---|---|---|---|---|
| | | Screening evaluation | Study drug administration | Clinical assessment | Engraftment | Research<br>lab samples | Survey |
| Scr | eening Visit | Х | | Х | | | |
| Pre-conditioning | | | х | | | Х | Х |
| Transplant (Day 0) | | | | х | | х | |
| | Day 7 | | | X | | x | |
| | Day 14 | | | Х | | Х | |
| | Day 21 | | | Х | | | |
| | Day 28 | | | X | X | X | |
| | Day 35 | | | Х | | | |
| | Day 42 | | | Х | | | |
| | Day 49 | | | Х | | | |
| | Day 50 | | х | | | | |
| | Day 56 | | | Х | | X | |
| Post-Transplant | Day 63 | | | Х | | | |
| | Day 70 | | | Х | | | |
| | Day 77 | | | Х | | | |
| | Day 84 | | | Х | | | |
| | Day 91 | | | Х | | Х | |
| | Day 98 | | | Х | | | Х |
| | Day 100 | | x | | | | |
| | 4 months | | | Х | | x | |
| | Day 160 | | x | | | | |
| | 6 months | | | Х | | Х | Х |
| | 9 months | | | Х | | Х | |
| | 12 months | | | Х | | Х | Х |
| | 18 months | | | Х | | | |
| | 24 months | | | Х | | | X |

<sup>\*</sup> In addition to the research blood samples outlined above, you will have the option to allow collection of research samples from your marrow any time a bone marrow test is being done for your routine care (for example, at day 30 and 90, at 1 year, or if your blood counts are abnormal). The research sample would be collected during your already planned bone marrow biopsy (meaning that you would not need to undergo a separate bone marrow biopsy procedure for this). As these are optional, you can elect to either allow them or not.

# How long would you stay in this study?

If you join this study, we think you would stay in this study for about 2 years after transplant.

Doctors could decide that you should stop taking the study drug (ustekinumab or placebo) but continue with study follow up assessments. This would happen if:

- They think it is in your best interest not to continue in the study.
- You have unacceptable toxicity from the treatment.
- You are not able or willing to follow study procedures.
- You develop severe acute GVHD.
- Your disease returns after transplant (relapse).

Under certain circumstances, doctors could decide that you should stop taking the study drug and discontinue participation from all follow up procedures. This would happen if:

- You decide to withdraw from the study.
- The whole study is stopped.

If you decide to withdraw from the study, there is no penalty or loss of benefits in your routine medical care or any other benefit(s) that you would otherwise be entitled to receive.

If you withdraw from the study for any reason, previously collected information would remain in the study records and would be included in the analysis of results. This information could not be removed from the study records.

# What are the side effects (risks)?

In this part of the consent form, we describe the side effects we expect from the tests and treatments in this study. If you join this study, we would tell you if we discover new side effects that could affect you.

Tacrolimus and methotrexate are standard medications used to prevent GVHD but they will suppress your immune system and increase the risk of infection. Infection, severe allergic reactions, and other side effects can lead to death. The side effects described below are seen in patients undergoing stem cell transplants, although their occurrence and severity will vary from person to person. With any medication or combination of medications, there may be complications or other side effects that we do not know about. Some side effects may require that we decrease the dose of these medications or hold the medication. Your doctor (attending physician) may suggest that you take certain medications to reduce some of the side effects.

#### Side effects of Tacrolimus:

• Decline in liver or kidney function that, if severe, may require the use of an artificial kidney machine (hemodialysis)

- Pain in the hands and feet or shaking of the hands (tremor)
- Loss of appetite, nausea, vomiting, or diarrhea
- Breakdown of red blood cells (hemolysis)
- Back pain
- Skin rash or itchy skin (pruritus)
- Loss of magnesium or increased levels of potassium or glucose
- High blood pressure (hypertension)
- Confusion, headache, and, infrequently, seizures
- Difficulty sleeping
- Blurred vision or sensitivity to bright light
- Increased fats (hyperlipidemia) in blood
- Posterior Reversible Encephalopathy Syndrome (PRES), swelling of the brain that may cause headache, seizures, confusion or loss of eyesight.

# **Side effects of Methotrexate:**

- Sores in the mouth or on the lips (mucositis)
- Slow recovery of blood cells after transplant
- Decline in liver function
- Nausea and vomiting

Many of these side effects go away once the medications are stopped, but sometimes side effects are very severe and long lasting. There also is a risk of death. We will do everything possible to lessen these side effects. If you want to read more about these medications, please ask the doctor (attending physician) or pharmacist for more information.

# Potential Discomforts, Side Effects and Risks Associated with Ustekinumab

The possible discomforts, side effects and risks related to Ustekinumab treatment are not all known. Most side effects are not serious. Some may be serious and may require treatment or additional testing. This section describes how frequently side effects occurred in subjects who were treated with Ustekinumab. In this section, the following terms are used:

- Very common: affects more than 1 user in 10
- Common: affects 1 to 10 users in 100
- Uncommon: affects 1 to 10 users in 1,000
- Rare: affects 1 to 10 users in 10,000
- Very rare: affects less than 1 in 10,000 users

#### **Very Common:**

• None.

#### Common:

- Infection of the throat, airway or sinus
- sore throat
- feeling tired
- redness and pain at drug injection site
- back, joint or muscle pain
- vomiting

- Headache
- dizziness
- diarrhea
- nausea
- itchiness

#### Uncommon:

- Swelling, itching, hardness, bleeding, bruising and irritation where the injection is given.
- Shingles (a painful rash)
- Depression
- Inflammation of tissue under the skin. Signs include warmth, swelling, redness and pain
- nasal congestion
- a form of psoriasis with raised bumps on the skin that are filled with pus
- Allergic reactions including rash or raised, itchy bumps
- tooth infections
- acne
- feeling weak
- vaginal yeast infection
- chest infection

#### Rare:

- Serious allergic reactions, which could be life-threatening (including low blood pressure, trouble breathing, swollen face, lips, mouth and/or throat)
- A form of psoriasis with redness and scaling of a much larger area of your skin or your entire body (erythrodermic psoriasis)
- In rare cases, symptoms such as cough, shortness of breath, and fever may also be a sign of an allergic lung reaction to Ustekinumab
- Inflammation of small blood vessels, which can lead to a skin rash with small red or purple bumps, fever or joint pain (vasculitis).

#### Very Rare:

• None.

# Infections

Ustekinumab is a drug that may change how your body fights infections. Serious infections requiring hospitalization for medical observation and /or treatment have been seen in Ustekinumab studies. Some of these infections have also been life threatening.

Tell your study doctor if you have a new infection, if an infection keeps coming back, or if you have any signs of infection such as:

- fever
- chills
- headache
- coughing
- congestion
- chest tightness
- shortness of breath
- flu-like symptoms
- nausea
- vomiting
- diarrhea
- increased frequency or burning while passing urine
- redness warmth, tenderness or swelling of skin or joint
- cold sores
- new or worsening of pain in any location
- weight loss
- tiredness
- night sweats

It is unknown if Ustekinumab may stop you from developing a fever if you do have an infection, and therefore hide that you have one.

Fungal infections have been reported in subjects taking Ustekinumab. Some of these fungal infections can be serious and involve internal organs. You should find out from your study doctor which fungal infections are common where you live or travel and what symptoms they cause. Tell your study doctor and family physician right away if you develop symptoms of such illnesses.

Subjects who receive Ustekinumab may also be at a greater risk for certain serious infections such as tuberculosis. Tell your study doctor if you have ever had tuberculosis or anybody in your family has ever had tuberculosis or if you come in contact with someone who has tuberculosis. You will have a screening test for tuberculosis before you start the study treatment. Tell your study doctor if you develop:

- a cough that does not go away
- coughing up blood
- shortness of breath
- fever
- night sweats
- weight loss

#### Cancer

Cancers have been reported in subjects who have received Ustekinumab but it is unknown whether taking Ustekinumab has increased their risk for developing cancer. Because Ustekinumab may suppress your immune system, it is possible that it may increase your risk of developing cancer, including skin cancers. Subjects who have been diagnosed with psoriasis have a higher chance of developing skin cancers. Tell your doctor if you have any new or changing skin lesions.

It is known that people who have had inflammatory diseases (such as, Crohn's disease, Rheumatoid Arthritis, Ulcerative Colitis etc.) for a long time and who use immunosuppressive therapies (such as, azathioprine, methotrexate etc.) for a long time have a higher risk of developing cancer. These people get cancer of the lymph nodes more often than other people.

# Infusion Reactions, Injection Site Reactions and Allergic Reactions

Ustekinumab may cause an allergic reaction in some subjects. These reactions are usually mild to moderate. Your body might have a reaction during or shortly following an infusion of Ustekinumab into the vein. This is called an infusion reaction and these reactions are usually mild to moderate. They are managed by slowing the infusion or by giving you medication. The following can be symptoms of an infusion reaction or an allergic reaction:

- fever
- chills
- hives
- rash
- swelling
- itching
- headache
- flushing
- nausea
- light-headedness
- chest pain or tightness
- wheezing
- difficulty breathing or swallowing
- decrease or increase in blood pressure
- anaphylaxis (life threatening allergic reaction)

Serious allergic reactions have been reported in subjects taking Ustekinumab and can be life threatening. If this happens during the infusion, the infusion will be stopped. Signs of a serious allergic reaction include skin rash, swollen face, mouth, lips, and/or throat, and trouble breathing. Tell your doctor or get emergency medical help right away if you have an allergic reaction. If you experience a serious reaction to an injection or an infusion, you will not receive any more study treatments.

If you have an infusion reaction or an allergic reaction at the doctor's office, additional necessary treatment will be provided immediately. Your study doctor may give you an antihistamine (medication used to treat allergic symptoms such as hay fever) or other medications used for treating an allergy. Antihistamines can make you sleepy, so please use caution when driving a car or operating machinery.

Another type of allergic reaction has occurred in some subjects 1-14 days after receiving some similar medications. The symptoms of this type of allergic reaction may include fever, rash, muscle aches and joint pain.

#### **Antibodies to Ustekinumab**

Sometimes the body can make special antibodies that may increase the risk of an allergic reaction to either Ustekinumab or other antibody medicines. If you have an allergic reaction, you may not be able to have these types of medications in the future. You should always tell your doctors that you have been treated with human antibodies in this study.

#### Cardiac and Vascular

Heart attacks and strokes have been reported in subjects who have received Ustekinumab. These events have rarely resulted in death. It is unknown whether taking Ustekinumab increases your risk for developing these events.

People who have psoriasis, and certain other inflammatory diseases, have a higher risk of having heart attacks. These people have heart attacks more often than other people. Seek medical care immediately if you develop;

- chest pain or discomfort
- trouble breathing
- irregular heartbeats
- dizziness
- loss of balance
- new numbness or weakness
- visual or speech changes

#### **Vaccination**

Vaccines are made to help protect people from certain illnesses. Some vaccines are made from live bacteria or live viruses. You cannot receive most kinds of live vaccines (for example, FluMist<sup>TM</sup>, varicella) during the study or for 3 months after the last study injection. Another kind of live vaccine is BCG, which is a vaccine against tuberculosis. You cannot receive a BCG vaccine during this study or for 12 months after the last study injection. You could get sick from these kinds of vaccines while on Ustekinumab. If you do get a live vaccination during this study, you must tell your study doctor immediately.

Tell your study doctor if anyone living in your home needs a live vaccine. Some viruses used in live vaccines can spread from a close contact (someone living in your home) to people with a weakened immune system.

Other kinds of vaccines, like tetanus and flu shots, and COVID vaccines that are not live, are allowed. It is not known if Ustekinumab may interfere with them from working. Tell your study doctor before getting any vaccine while you are in this study.

# Allergy Immunotherapy (Allergy Injections)

Tell your study doctor if you have ever had or are now getting allergy injections. Ustekinumab may affect your response to allergy injections.

#### Other Risks

Two cases of a very rare disease of the brain, known as PRES (posterior reversible encephalopathy syndrome), have been reported in clinical trials with Ustekinumab. Cases have also been reported in post marketing experience in patients with psoriasis, psoriatic arthritis and Crohn's disease. PRES is generally reversible and is not caused by an infection. It is unknown whether taking Ustekinumab increases your risk of developing PRES. Symptoms of this condition are:

- headache
- seizures
- confusion
- loss of eyesight

Tell your study doctor if you experience any of these symptoms. There may be other discomforts or risks to you from this study that are not yet known. Your study doctor and staff will ask you about any side effects you may have at every visit. If you have any problems, you should let your study doctor know right away.

Tell your doctors or dentist that you are or have been in a study where anti IL-12 and anti IL-23 is the study drug. This is important if you have any surgery, dental procedures, or receive treatment for any other medical condition.

# What about birth control and pregnancy during the study?

The effect of Ustekinumab on human sperm or unborn babies is not known.

Pregnant women and women who are making breast milk to feed infants cannot participate in this study. Female subjects must have a blood test when beginning this study that shows they are not pregnant.

It is very important that women taking part in this study do not become pregnant while taking part in this study. It is very important that men taking part in this study do not get a woman pregnant while taking part in this study.

During this study and for at least 15 weeks after the last dose of study drug, women of childbearing potential and men must use proven birth control methods. Your study doctor will discuss effective birth control methods with you.

Examples of birth control methods include:

- Oral birth control pills
- Birth control patch
- Implanted (injectable contraceptive hormones or mechanical products such as intrauterine device)
- Barrier methods (diaphragm, condoms, spermicidal)
- Tubal ligation or vasectomy
- Abstinence (no sexual intercourse)

If you think that you have become pregnant or may have fathered a child while taking part in the study, tell your study doctor immediately. You should also notify your childbirth doctor that the mother/father received an experimental drug (Ustekinumab).

If you are a female study subject and you become pregnant during your participation in this study, your treatment with study drug will be stopped and you may be withdrawn from some of the study procedures but not from follow-up by your study doctor. The study doctor will ask for your permission to stay in contact with you throughout the length of the pregnancy.

It's also important that you tell your baby's doctor and other health care professionals that you received treatment with Ustekinumab while pregnant, because a 6-month waiting period following birth may be recommended before the administration of a live vaccine (like BCG and rotavirus) to the baby.

If you are a female study subject, you must not donate eggs during the study and for at least 15 weeks after your last dose of study drug.

If you are a male study subject, and you father a child during your participation in this study, the study doctor will ask for your partner's permission to stay in contact with her throughout the length of the pregnancy.

If you are a male study subject, you must not donate sperm during the study and for at least 15 weeks after your last dose of study drug.

The long-term effects of the study treatment on fertility are unknown. This means that it is unknown if treatment with these medications will affect your ability to have children in the future.

# **Tuberculosis testing**

You will be tested with a tuberculosis screening blood test prior to joining the study. If your test shows you likely have tuberculosis, you would not be eligible for the study, and your doctor would talk to you about the appropriate next steps in your medical care for tuberculosis.

#### **Additional Risks**

Risks of blood draws include fainting, dizziness, mild bleeding or bruising, and the risk of infection at the needle site.

To check for GVHD, it may be necessary to get a biopsy (small piece of tissue) from your skin, stomach or liver. The primary side effects related to this procedure are pain, bleeding or bruising the biopsy site. Infrequently, you may develop an infection at the biopsy site.

It is possible that completing the questionnaires may cause fatigue or you may experience emotional distress.

There is a risk of loss of confidentiality of your information. Results of your genetic tests may be released by accident. This risk is very low, because we keep your personal information private. If your results become known, you may have problems with family members or insurance.

You will read more about the protection of your information later in this form. Please ask the study doctor or study staff if you would like to know more about how your information will be protected while you are in this study.

### What are the benefits?

We do not know if this study would help you. We are testing ustekinumab to see its effects on people at risk of developing GVHD after stem cell transplant. You might get better if you receive the study drug (ustekinumab or placebo), but your condition could stay the same or even get worse. We hope the information from this study will help other people undergoing stem cell transplants in the future.

### You have other choices besides this study.

You do not have to join this study. You are free to say "yes" or "no". Your regular medical care would not change if you decide to say "no".

You have other choices for treatment. Each of these choices has risks and benefits. You should talk to your doctor or healthcare provider about these choices.

Other choices include: treatment with tacrolimus and methotrexate alone, participation in another research study, or using other available regimens for preventing GVHD.

Enrollment in this study may exclude you from other research studies.

# Protecting Privacy as an Individual and the Confidentiality of Personal Information

If you join this study, some people or organizations might need to look at your medical records and research records for quality assurance or data analysis. They include:

- Researchers involved with this study.
- Janssen, Johnson and Johnson and their agents.
- Institutional Review Boards (IRB), including the Fred Hutchinson Cancer Center IRB. An IRB is a group that reviews the study to protect the rights and welfare of research participants.
- Fred Hutchinson Cancer Center, University of Washington, and Seattle Cancer Care Alliance.
- Office for Human Research Protections, Food and Drug Administration, and other regulatory agencies as required.

We will do our best to keep personal information confidential. But we cannot guarantee total confidentiality. Personal information may be given out if required by law. For example, workplace safety rules may require health workers to contact you about lab tests. Or a court may order study information to be disclosed. Such cases are rare.

We will not use personal information in any reports about this study, such as journal articles or presentations at scientific meetings.

If you join this study, information about your participation would be made part of your permanent medical record. This information would include a copy of this consent form. If an insurance company or employer or anyone else were authorized to see your medical record, they would see a copy of this consent form.

This research is covered by a Certificate of Confidentiality from the U.S. government. This Certificate helps protect the confidentiality of information about people who join this study. If you join the study, the Certificate means that generally we would not have to give out identifying information about you even if we were asked to by a court of law. We would use the Certificate to resist any demands for identifying information.

We could not use the Certificate to withhold research information if you give written consent to give it to an insurer, employer, or other person.

This protection has some limits. We would voluntarily provide the information:

- To a member of the federal government who needs it in order to audit or evaluate the research.
- To the funding agency and groups involved in the research, if they need the information to make sure the research is being done correctly.
- To the federal Food and Drug Administration (FDA), if required by the FDA.

- To someone who is accused of a crime, if he or she believes that our research records could be used for defense.
- To authorities, if we learn of child abuse, elder abuse, or if participants might harm themselves or others.

# How is my genetic information protected?

A federal law called the Genetic Information Nondiscrimination Act (GINA) helps protect genetic information about people who join research studies.

GINA restricts access to genetic information so that it cannot be used for health insurance coverage decisions. GINA prevents health insurance companies or group health plans from:

- Asking for genetic information obtained in research studies, or
- Using genetic information when making decisions regarding your eligibility or premiums

GINA *does not* help or protect against genetic discrimination by companies that sell life, disability or long-term care insurance.

# Would we pay you if you join this study?

There is no payment for being in this study.

# Would you have extra costs if you join this study?

If you join this study, the study-specific treatments and study-required assessments (for example, extra blood samples drawn for research, pregnancy tests, or questionnaires) will be paid for by the study budget and not billed to you or your insurance provider.

In contrast, as is true if you were not taking part in this study, you or your insurance provider is responsible for the routine aspects of your medical care that are not direct components of this study (medications, tests, clinic and hospital visits as part of your routine care as a transplant recipient).

However, there are possible additional charges to you or your insurance provider listed here below. Your insurance company might pay these costs, but some insurance policies do not cover these costs. We could help find out whether your insurance company would cover these costs.

#### The extra costs are:

• Cost of tests that are given more often than usual.

- Cost of people and equipment to give the study drug (ustekinumab or placebo). There is no charge for the study drug itself.
- Cost of any other medical care needed because of this study.

# What if you get sick or hurt after you join this study?

For a life-threatening problem, call 911 right away or seek help immediately. Contact your study doctor when the medical emergency is over or as soon as you can.

For all other medical problems or illness related to this research, immediately contact Dr. Lee at 206-667-5160. They will treat you or refer you for treatment. You or your health insurance will have to pay for the treatment. There are no funds to pay you for a research-related injury, added medical costs, loss of a job, or other costs to you or your family. State or national law may give you rights to seek payment for some of these expenses. You do not waive any right to seek payment by signing this consent form.

You or your insurer will be billed for treatment of problems or complications that result from your condition or from standard clinical care.

You would not lose any legal right to seek payment for treatment if you sign this form.

# What will my information and/or tissue samples be used for?

Your information and samples will be used for the purposes of this study.

Your samples might help researchers develop new products. This research could be done by for-profit companies. There is no plan to share with you any revenue generated from products developed using your tissue samples.

During this study, we do not expect any research test results that would affect your care, so we do not plan to return results to you.

In addition, by agreeing to participate in this study, your information or samples could be used for future research studies or sent to other investigators for future research studies without additional consent from you. These future research studies will be reviewed by an oversight group known as an institutional review board if required by law. The information that identifies you will first be removed from your information or samples.

# **DNA** sequencing

Each cell in your body contains thousands of genes which control the activity of cells. Researchers can now examine all the genes in these cells. How genes control cell function is encoded in your DNA. To study genes that contribute to graft vs. host disease or a related disorder, we are requesting permission to sequence (read)

your DNA. This may be small regions of the DNA or the entire DNA molecule (whole genome sequencing). This work is generally called genetic research or genetic studies. Sometimes samples are used for genetic research about traits that are passed on in families (inherited). There are other genetic changes that are not inherited or passed on in families but are related to the disease process. These genes may only be found in blood, bone marrow, or other tissue affected by the disease. Sometimes we need to compare the genetic sequence in skin cells with blood, marrow, or cells from other tissue to determine which genetic sequence changes are related to your disease. As new technology advances, we may sequence your DNA sample in the future in a way that we cannot predict today.

This type of testing can provide useful information to researchers. It can also present risks if the test results became known to others, for example you could have problems with family members or insurance companies. There is also a risk that these test results could be combined with other genetic information to identify you.

# We invite you to donate samples for other research.

After we do tests on samples in this study, some samples may be left over. We invite you to donate the leftover samples for future research. This may include genetic research.

If you join this study, you would not have to donate samples for future research. You would be free to say "yes" or "no." Regular medical care would not change if you say "no."

If you donate samples, they would be stored in a secure location. If we want to use your samples for other research or share it with other scientists for research, an ethics review committee (IRB) would review the request. The IRB would decide if we need to ask you for permission to do the research.

Your donated samples would be used only for research. This research could be done by for-profit companies. Researchers would not report their results to you or your doctors. The research results would not be included in medical records. The results would not affect your medical care.

Research with samples might help develop new products. If these products make money, there is no plan to share the money with the participants who donate the tissue.

If you donate samples for research, you could withdraw the donation at any time by calling Dr. Lee at 206-667-5160. You would have no penalty for withdrawing the donation, and regular medical care would not change. We could not return donated samples, but we might be able to destroy the donated samples. We could not destroy samples if it is stored or shared without any label saying who donated it. In this case, it could still be used for research.

# Your rights

- You do not have to join this study. You are free to say "yes" or "no".
- If you get sick or hurt in this study, you do not lose any of your legal rights to seek payment by signing this form.
- During the study, we might learn new information that you need to know. For example, some information may affect your health or well-being. Other information might make you change your mind about being in this study. If we learn these kinds of information, we would tell you.
- If you join this study, you would not have to stay in it. You could stop at any time (even before you start). Your regular medical care would not change. You would have no penalty for stopping, but it would be better not to join the study if you think that you would change your mind later.

A description of this clinical trial will be available on *http://www.ClinicalTrials.gov*, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# Your responsibilities

If you join this study, you would have some responsibilities.

- Follow the schedule of study visits and procedures.
- Take study medications as directed.
- Prevent pregnancy.
- Tell us about side effects.

#### For more information

If you have questions or concerns about this study, you can talk to your doctor anytime. Other people you could talk to are listed below.

| If you have questions about: | Call: |
|---|---|
| This study (including complaints and requests for information) | (206) 667-5160 (Dr. Stephanie Lee)<br>(206) 667-4160 (Research Coordinator) |
| If you get sick or hurt in this study | (206) 667-5160 (Dr. Lee) |
| Your rights as a research participant | 206-667-5900 or email irodirector@fredhutch.org<br>(Director of Institutional Review Office, Fred<br>Hutchinson Cancer Center) |
| Your bills and health insurance coverage | (206) 606-6226 or toll free at (800) 804-8824 |

# Emergency number (24 hours): (206) 598-8902

Read each question and think about your choice. When you decide on each question, please circle **YES** or **NO**.

Do you agree to give extra bone marrow for research when bone marrow sampling is performed for clinical purposes?

(circle one)

YES NO

Do you agree to donate your leftover samples for future studies of transplant complications?

(circle one)

YES NO

#### Genetic research:

As part of this study we may want to put your genetic information into shared databases in the future. Or we may be required to put your genetic information into a

Fred Hutch IRB Approved 5/3/2023

protected database when results of studies using your genetic information are published in a scientific journal.

Several genetic databases are available to help researchers understand different diseases. These databases contain DNA information and other data helpful to study diseases. DNA comes from cells in your body and contains all your genetic information. All of your personal information would be removed. Your name, address, etc. will not be in the database. Only genetic information and information about your condition will be sent to the database.

Your information may benefit future research.

There is a small risk that your genetic information could be matched against other genetic databases to get your name. Once we release your data to the central database we are no longer in control of the information.

| Is it OK if we send your genetic information to one or more databases? (circle one) | | | |
|---|---|---|---|
| YES | NO | Initials: | Date: |

# **Signatures**

Please sign below if you:

- have read this form (or had it read to you);
- had the opportunity to ask any questions you have;
- had the opportunity to discuss the research with the person obtaining consent; and
- agree to participate in this study.

Current consent version date: 12 September 2022 Previous consent version date: 14 April 2022

| Participant: | | |
|---|---|---|
| Printed Name | Signature | Date |
| below to indicate you a<br>apparent understanding | erpreter or impartial witness during attest to the accuracy of the presentag of and willingness to participate in | ation and the participant's |
| Impartial Witness or Inte | rpreter: | |
| Printed Name | Signature | Date |
| Researcher's statement | | |
| | ch study, including procedures and<br>he signed consent form will be give | <del>-</del> |
| Person obtaining consent | signature: | |
| Printed Name | Signature | Date |
| Protocol: RG1005588 | | |